CLINICAL TRIAL: NCT02224781
Title: DREAMseq (Doublet, Randomized Evaluation in Advanced Melanoma Sequencing) a Phase III Trial
Brief Title: Dabrafenib and Trametinib Followed by Ipilimumab and Nivolumab or Ipilimumab and Nivolumab Followed by Dabrafenib and Trametinib in Treating Patients With Stage III-IV BRAFV600 Melanoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01747; NCI-2014-01747 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA6134 (Other: ECOG-ACRIN Cancer Research Group); EA6134 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2014-08-22; First posted 2014-08-25 (Estimated); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Melanoma; Recurrent Melanoma; Unresectable Melanoma
MeSH Terms: conditions — Melanoma | interventions — Specimen Handling; dabrafenib; Ipilimumab; CTLA-4 Antigen; Nivolumab; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (immunotherapy) (Experimental): IMMUNOTHERAPY INDUCTION (CYCLES 1-2): Patients receive nivolumab IV over 30-60 minutes and ipilimumab IV over 30-90 minutes on days 1 and 22. Treatment repeats every 6 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity.
  IMMUNOTHERAPY MAINTENANCE (CYCLES 3-14): Patients receive nivolumab IV over 30-60 minutes on days 1, 15, and 29. Treatment repeats every 6 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Upon disease progression (or before), patients re-register and cross over to Arm C.
  Patients also undergo CT, ECHO or MUGA, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Biological: Ipilimumab; Procedure: Multigated Acquisition Scan; Biological: Nivolumab; Other: Quality-of-Life Assessment
- Arm B (BRAF inhibitor therapy) (Experimental): Patients receive dabrafenib mesylate PO BID and trametinib dimethyl sulfoxide PO daily on days 1-42. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Upon disease progression (or before), patients re-register and cross over to Arm D.
  Patients also undergo CT, ECHO or MUGA, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dabrafenib Mesylate; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Other: Quality-of-Life Assessment; Drug: Trametinib Dimethyl Sulfoxide
- Arm C (BRAF inhibitor therapy) (Experimental): Patients receive dabrafenib mesylate PO BID and trametinib dimethyl sulfoxide PO daily on days 1-42. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Patients also undergo CT, ECHO or MUGA, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dabrafenib Mesylate; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Other: Quality-of-Life Assessment; Drug: Trametinib Dimethyl Sulfoxide
- Arm D (immunotherapy) (Experimental): IMMUNOTHERAPY INDUCTION (CYCLES 1-2): Patients receive nivolumab IV over 30-60 minutes and ipilimumab IV over 30-90 minutes on days 1 and 22. Treatment repeats every 6 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity.
  IMMUNOTHERAPY MAINTENANCE (CYCLES 3-14): Patients receive nivolumab IV over 30-60 minutes on days 1, 15, and 29. Treatment repeats every 6 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Patients also undergo CT, ECHO or MUGA, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Biological: Ipilimumab; Procedure: Multigated Acquisition Scan; Biological: Nivolumab; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Dabrafenib Mesylate — Given PO
  Other Names: Dabrafenib Methanesulfonate; GSK2118436 Methane Sulfonate Salt; GSK2118436B; Tafinlar
  Arms: Arm B (BRAF inhibitor therapy); Arm C (BRAF inhibitor therapy)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Arm A (immunotherapy); Arm D (immunotherapy)
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; MUGA; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm A (immunotherapy); Arm D (immunotherapy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Trametinib Dimethyl Sulfoxide — Given PO
  Other Names: Mekinist; Meqsel; Spexotras
  Arms: Arm B (BRAF inhibitor therapy); Arm C (BRAF inhibitor therapy)

SUMMARY:
This phase III trial studies how well initial treatment with ipilimumab and nivolumab followed by dabrafenib and trametinib works and compares it to initial treatment with dabrafenib and trametinib followed by ipilimumab and nivolumab in treating patients with stage III-IV melanoma that contains a mutation known as BRAFV600 and cannot be removed by surgery (unresectable). Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Dabrafenib and trametinib may block tumor growth by targeting the BRAFV600 gene. It is not yet known whether treating patients with ipilimumab and nivolumab followed by dabrafenib and trametinib is more effective than treatment with dabrafenib and trametinib followed by ipilimumab and nivolumab.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether initial treatment with either combination ipilimumab + nivolumab (with subsequent dabrafenib mesylate [dabrafenib] in combination with trametinib dimethyl sulfoxide [trametinib]) or dabrafenib in combination with trametinib (with subsequent ipilimumab + nivolumab) significantly improves 2 year overall survival (OS) in patients with unresectable stage III or stage IV BRAFV600 mutant melanoma.

SECONDARY CLINICAL OBJECTIVES:

I. To evaluate the impact of initial treatment on median OS and hazard ratio for death.

II. To determine whether initial treatment choice significantly improves 3 year OS.

III. To evaluate the anti-tumor activities (Response Evaluation Criteria in Solid Tumors [RECIST]-defined response rate, median progression-free survival [PFS]) and safety profiles of ipilimumab + nivolumab and dabrafenib-trametinib in a Cooperative Group trial of patients with V600 mutant melanoma.

IV. To evaluate the activity (RECIST-defined response rate, median PFS) and safety of dabrafenib + trametinib in patients who have had disease progression on ipilimumab + nivolumab and in comparison to its activity and safety in ipilimumab + nivolumab naive patients.

V. To evaluate the activity of ipilimumab + nivolumab (RECIST-defined response rate, median PFS) and safety in patients who have had disease progression on dabrafenib + trametinib and in comparison to its activity and safety in dabrafenib + trametinib naive patients.

VI. To assess the feasibility of crossover to the alternative treatment strategy (percentage of patients who are able to crossover from one arm to the other and complete at least an initial course [12 weeks] of treatment after cross-over without intervening symptomatic disease progression or treatment limiting toxicity).

SECONDARY LABORATORY OBJECTIVES:

I. Association of inherited variation with immune mediated adverse events and response to ipilimumab + nivolumab.

Ia. To determine the association of inherited genetic variation and immune-associated adverse events in patients with metastatic melanoma treated with ipilimumab containing regimens by completing candidate-based gene and pathway analyses of genes involved in lymphocyte activation, cytokines, cytokine receptors and within the major histocompatibility complex (MHC) region and an agnostic genome-wide single nucleotide polymorphism (SNP)-based approach; Ib. To investigate the association between inherited genetics and survival in patients with metastatic melanoma treated with ipilimumab containing regimens by completing candidate-based gene and pathway analyses of genes involved in lymphocyte activation, cytokines profile, cytokine receptors and within the MHC region and an agnostic genome-wide SNP-based approach; Ic. To replicate genomic markers identified in the above aims in an independent sample set of patients treated with ipilimumab containing regimens and preliminarily characterize their potential functional role by completing replication of variation as associated with immune-related adverse events (irAEs) and survival and bio-informatic assessment of genomic markers.

II. To determine the utility of circulating BRAF levels in determining the response and resistance to either BRAF/MEK directed and/or combination immunotherapy in patients with BRAF mutant melanoma.

IIa. To determine if changes in blood BRAF levels utilizing peripheral blood BRAFV600 mutational testing in patients with stage IV BRAF mutant melanoma correlate with response and resistance to combination BRAF/MEK directed therapy; IIb. To determine if changes in blood BRAF levels utilizing peripheral blood BRAFV600 mutational testing in patients with stage IV BRAF mutant melanoma correlate with response and resistance to combination immunotherapy; IIc. To compare the kinetics of peripheral blood BRAFV600 levels during response and resistance in groups of patients receiving BRAF targeted therapy or combination immunotherapy as initial therapy; IId. To compare the kinetics of peripheral blood BRAFV600 levels during response and resistance to combination BRAF targeted therapy or combination immunotherapy in individual patients (initial treatment versus [vs] crossover treatment).

SECONDARY PATIENT REPORTED OUTCOMES OBJECTIVES:

I. To evaluate differences in overall health between initial treatment arms (dabrafenib + trametinib vs. ipilimumab + nivolumab immunotherapy) at 2 years, accounting for toxicities and overall survival. (Primary) II. To assess differences in overall function over 2 years between initial treatment with dabrafenib + trametinib vs. ipilimumab + nivolumab. (Secondary) III. To document the effects of treatment crossover and treatment administration sequence on symptom burden and overall function. (Secondary) IIIa. To compare differences in function and symptoms by treatment sequence for ipilimumab + nivolumab (arm A vs. D), and dabrafenib + trametinib, (arm B vs. C) at baseline, 6 weeks, 12 weeks, and 6 months after the initiation of each treatment; IIIb. To describe the frequency and severity of treatment toxicities at baseline, 6 weeks, 12 weeks, and 6 months after initiation of each treatment.

EXPLORATORY TOBACCO USE OBJECTIVES:

I. To determine the effects of tobacco, operationalized as combustible tobacco (1a), other forms of tobacco (1b), and environmental tobacco exposure (ETS) (1c) on provider-reported cancer-treatment toxicity (adverse events [both clinical and hematologic] and dose modifications).

II. To determine the effects of tobacco on patient-reported physical symptoms and psychological symptoms.

III. To examine quitting behaviors and behavioral counseling/support and cessation medication utilization.

IV. To explore the effect of tobacco use and exposure on treatment duration, relative dose intensity, and therapeutic benefit.

EXPLORATORY CORRELATIVE OBJECTIVES:

I. To assess serum based biomarkers of efficacy and adverse events due to treatment with immune checkpoint inhibitors.

II. To monitor tumor response by comparing changes in circulating cell-free mutant tumor deoxyribonucleic acid (DNA) (ctDNA) as a readout of tumor burden (a) at week 12 relative to baseline before treatment in responders and non-responders; (b) before and during immunosuppressive treatment to control irAEs.

III. To monitor organ-specific adverse events (irAEs) using circulating cell-free, tissue-specific methylated DNA (cmeDNA) as a readout of tissue-specific toxicity (a) at the time of grade 3-4 irAE relative to baseline and control patients without irAEs; (b) during immunosuppressive treatment for irAEs.

OUTLINE: Patients are randomized to 1 of 2 treatment arms (Arm A or Arm B).

ARM A:

IMMUNOTHERAPY INDUCTION (CYCLES 1-2): Patients receive nivolumab intravenously (IV) over 30-60 minutes and ipilimumab IV over 30-90 minutes on days 1 and 22. Treatment repeats every 6 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity.

IMMUNOTHERAPY MAINTENANCE (CYCLES 3-14): Patients receive nivolumab IV over 30-60 minutes on days 1, 15, and 29. Treatment repeats every 6 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Upon disease progression (or before), patients re-register and cross over to Arm C.

ARM C: Patients receive dabrafenib mesylate orally (PO) twice daily (BID) and trametinib dimethyl sulfoxide PO daily on days 1-42. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive dabrafenib mesylate PO BID and trametinib dimethyl sulfoxide PO daily on days 1-42. Cycles repeat every 6 weeks in the absence of disease progression or unacceptable toxicity. Upon disease progression (or before), patients re-register and cross over to Arm D.

ARM D:

IMMUNOTHERAPY INDUCTION (CYCLES 1-2): Patients receive nivolumab IV over 30-60 minutes and ipilimumab IV over 30-90 minutes on days 1 and 22. Treatment repeats every 6 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity.

IMMUNOTHERAPY MAINTENANCE (CYCLES 3-14): Patients receive nivolumab IV over 30-60 minutes on days 1, 15, and 29. Treatment repeats every 6 weeks for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

All patients also undergo computed tomography (CT), echocardiography (ECHO) or multigated acquisition scan (MUGA), and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of dabrafenib or dabrafenib + trametinib or nivolumab or nivolumab + ipilimumab therapy in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status: 0 or 1
* Women must not be pregnant or breast-feeding, as the effects of ipilimumab + nivolumab or dabrafenib + trametinib on the developing human fetus are unknown

  * All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
  * A female of childbearing potential is anyone, regardless of whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* The effects of dabrafenib and trametinib or ipilimumab and nivolumab on the developing human fetus are unknown; furthermore, dabrafenib has been reported to interfere with the effect of hormone based oral contraceptives; for this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and sexually active males must agree to use at least two other accepted and effective methods of contraception and/or to abstain from sexual intercourse for the duration of their participation in the study, and for at least 4 weeks after treatment with dabrafenib or for 4 months after dabrafenib in combination with trametinib; women of child-bearing potential must use at least two other accepted and effective methods of contraception and/or to abstain from sexual intercourse for at least 5 months after the last dose of nivolumab and/or ipilimumab. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Patients must have unresectable stage III or stage IV disease
* Patients must have measurable disease; all sites of disease must be evaluated within 4 weeks prior to randomization
* Patients must have histological or cytological confirmation of melanoma that is metastatic or unresectable and clearly progressive

  * NOTE: Any patient with BRAF V600 mutant melanoma (whether cutaneous, acral or mucosal primary) who meets the eligibility criteria is eligible for participation in this trial; patients with uveal melanoma are not eligible for this trial
* Patients must have BRAF V600 mutation, identified by a Food and Drug Administration (FDA)-approved test at a Clinical Laboratory Improvement Act (CLIA)-certified lab; if test at CLIA-certified lab used a non-FDA approved method, information about the assay must be provided (FDA approved tests for BRAF V600 mutations in melanoma include: THxID BRAF Detection Kit and Cobas 4800 BRAF V600 Mutation Test, Foundation Medicine); prompt information on tumor BRAF mutation status can also be obtained via Novartis "knowNow" Program
* Patients may have had prior systemic therapy in the adjuvant setting; however this adjuvant treatment must not have included a CTLA4 or PD1 pathway blocking antibody or a BRAF/MEK inhibitor. Also, patients may not have had any prior systemic treatment for advanced (measurable metastatic) disease
* Patients must have discontinued chemotherapy, immunotherapy or other investigational agents used in the adjuvant setting >= 4 weeks prior to entering the study and recovered from adverse events due to those agents; mitomycin and nitrosoureas must have been discontinued at least 6 weeks prior to entering the study; patients must have discontinued radiation therapy >= 1 week prior to entering the study and recovered from any adverse events associated with treatment; prior surgery must be >= 2 weeks from registration and patients must be fully recovered from post-surgical complications
* Patients must not receive any other investigational agents while on study or within four weeks prior to registration
* Patients are ineligible if they have any currently known active and definitive central nervous system (CNS) metastases; patients who have treated brain metastases (with either surgical resection or stereotactic radiosurgery [SRS]) could be eligible; patients must not have taken any steroids =< 10 days prior to randomization for the purpose of managing their brain metastases; repeat imaging after SRS or surgical resection is not required so long as baseline magnetic resonance imaging (MRI) is within 4 weeks of registration; patients with multiple brain metastases treated with SRS (with [w] or without [w/o] whole-brain radiotherapy [WBRT]), are not an exclusion; patients with definitive CNS metastases treated with only WBRT are ineligible; patients with potential CNS metastases that are too small for treatment with either SRS or surgery (e.g. 1-2 mm) and/or are of uncertain etiology are potentially eligible, but need to be discussed with and approved by the study principal investigator (PI)
* Patients must not have other current malignancies, other than basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast; patients with other malignancies are eligible if they have been continuously disease-free for > 2 years prior to the time of registration
* White blood count >= 3,000/uL (obtained within 4 weeks prior to randomization)
* Absolute neutrophil count (ANC) >= 1,500/uL (obtained within 4 weeks prior to randomization)
* Platelet count >= 100,000/uL (obtained within 4 weeks prior to randomization)
* Hemoglobin > 8 g/dL (obtained within 4 weeks prior to randomization)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or serum creatinine clearance (CrCl) >= 40 ml/min (obtained within 4 weeks prior to randomization)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN (=< 5 x ULN for patients with documented liver metastases) (obtained within 4 weeks prior to randomization)
* Alkaline phosphatase =< 2 x ULN (=< 5 x ULN for patients with known liver involvement and =< 7 x ULN for patients with known bone involvement) (obtained within 4 weeks prior to randomization)
* Total bilirubin =< 1.5 x ULN except subjects with normal direct bilirubin or those with known Gilbert's syndrome (obtained within 4 weeks prior to randomization)
* Patients must not have any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), including but not limited to, ongoing or active infection requiring parenteral antibiotics on day 1, or psychiatric illness/social situations that would limit compliance with study requirements, interfere with subject's safety, or obtaining informed consent; therapeutic level dosing of warfarin can be used with close monitoring of prothrombin time (PT)/international normalized ratio (INR) by the site; exposure may be decreased due to enzyme induction when on treatment, thus warfarin dosing may need to be adjusted based upon PT/INR; consequently, when discontinuing dabrafenib, warfarin exposure may be increased and thus close monitoring via PT/INR and warfarin dose adjustments must be made as clinically appropriate; prophylactic low dose warfarin may be given to maintain central catheter patency
* Patients must not have a history of or evidence of cardiovascular risks including any of the following:

  * QT interval corrected for heart rate using the Bazett's formula (QTcB) >= 480 msec. at baseline
  * History of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within the past 24 weeks prior to registration
  * History prior to registration or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Left ventricular ejection fraction (LVEF) =< 45% on cardiac echocardiogram (echo) or multi gated acquisition scan (MUGA)
  * Intra-cardiac defibrillator
* Individuals who are known to be human immunodeficiency virus (HIV) infected are ineligible (note: HIV testing is not required for entry into the study)
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease; patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), should be evaluated for the presence of target organ involvement and potential need for systemic treatment; if no systemic immune suppression is deemed necessary they can be eligible
* The following medications or non-drug therapies are also prohibited while on treatment in this study:

  * Other anti-cancer therapies
  * Other investigational drugs
  * Patients taking any medications or substances that are strong inhibitors or inducers of CYP3A or CYP2C8 are ineligible
* Patients must not have history of retinal vein occlusion (RVO)
* Patients must not have evidence of interstitial lung disease or pneumonitis
* Patients must not have malabsorption, swallowing difficulty, or other conditions that would interfere with the ingestion or absorption of dabrafenib or trametinib
* STEP 2 (CROSSOVER ARMS): The patient must have met all eligibility criteria (except as detailed below) at the time of crossover

  * RECIST defined measurable disease is not required
  * Only prior systemic therapy as part of step 1 is allowed; patients who received allowed systemic therapy in the adjuvant setting prior to Step 1 and were eligible for Step 1 are not excluded from proceeding to Step 2 if they meet other eligibility criteria
  * Malabsorption, swallowing difficulty, or other conditions that would interfere with the ingestion or absorption of dabrafenib or trametinib, or history of retinal vein occlusion are acceptable for patients crossing over to Arm D (ipilimumab + nivolumab) treatment
  * History of autoimmune disease, excluding interstitial lung disease or pneumonitis, is allowed in patients crossing over to Arm C (dabrafenib/trametinib) therapy
  * Patients crossing over from Arm A (nivolumab/ipilimumab) to Arm C (dabrafenib/trametinib) who underwent surgery or SRS to CNS metastases need not be off of steroids to start treatment
  * There is no restriction on serum lactate dehydrogenase (LDH) at crossover
  * Patients with a history of cardiovascular risks that developed during step 1 of therapy should be discussed with study principal investigator (PI) at time of crossover
* STEP 2 (CROSSOVER ARMS): Patients randomized to Arm A on Step 1 must have melanoma that is metastatic and clearly progressive on Step 1 therapy prior to crossing over to Arm C

  * NOTE: Patients should (if possible) be at least 1 week from documented PD on Step 1 of current study. All sites of disease must be evaluated within 4 weeks prior to registration
* STEP 2 (CROSSOVER ARMS): Patients randomized to Arm B on Step 1 may cross over to Arm D at or prior to disease progression

  * NOTE: If possible, patients should wait to cross over until after the cycle with the next protocol-required imaging assessment is completed; all sites of disease must be evaluated within 4 weeks prior to Step 2 registration
  * NOTE: Patients should start Arm D treatment at least 1 week after stopping dabrafenib and trametinib, unless otherwise clinically indicated
  * NOTE: Baseline labs and QOL assessments should be completed, and patients should follow the Arm D schedule
* STEP 2 (CROSSOVER ARMS): Patients must have recovered from adverse events (toxicities resolved to grade 1 or less) of prior therapy; patients with immune related toxicities from ipilimumab + nivolumab may continue onto Step 2 even if still on steroids to control side effects, so long as toxicity has resolved to grade 1 or less
* STEP 2 (CROSSOVER ARMS): Patients must have discontinued radiation therapy prior to registering to Step 2 of the study and recovered from any adverse events associated with treatment; prior surgery must be >= 2 weeks from registration to Step 2 and patients must be fully recovered from post-surgical complications
* STEP 2 (CROSSOVER ARMS): Patients are ineligible if they have any currently active and definitive CNS metastases; patients who have treated brain metastases (with either surgical resection or stereotactic radiosurgery [SRS]) could be eligible to proceed; patients crossing over from Arm B (dabrafenib/trametinib) to Arm D (nivolumab [nivo]/ipilimumab [ipi]) must not have taken any steroids =< 10 days prior to Step 2 registration for the purpose of managing their brain metastases; patients with only whole brain irradiation for treatment of CNS metastases are ineligible; patients with definitive CNS metastases treated with only WBRT are ineligible; patients with potential CNS metastases that are too small for treatment with either SRS or surgery (e.g. 1-2 mm) and/or are of uncertain etiology are potentially eligible, but need to be discussed with and approved by the study PI
* STEP 2 (CROSSOVER ARMS): Patients must not have other current malignancies
* STEP 2 (CROSSOVER ARMS): Women must not be pregnant or breast-feeding, as the effects of ipilimumab + nivolumab or dabrafenib + trametinib on the developing human fetus are unknown; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to Step 2 crossover to rule out pregnancy; a female of childbearing potential is anyone, regardless of whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months
* STEP 2 (CROSSOVER ARMS): The effects of dabrafenib and trametinib or ipilimumab and nivolumab on the developing human fetus are unknown; furthermore, dabrafenib has been reported to interfere with the effect of hormone based oral contraceptives; for this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and sexually active males must agree to continue to use the same contraception requirements as on Step 1 of this study (i.e.: use at least two other accepted and effective methods of contraception and/or to abstain from sexual intercourse for the duration of their participation in the study, and for at least 4 weeks after treatment with dabrafenib or for 4 months after dabrafenib in combination with trametinib; women of child-bearing potential must use at least two other accepted and effective methods of contraception and/or to abstain from sexual intercourse for at least 5 months after the last dose of nivolumab and/or ipilimumab. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2026-09-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) rate | The time from randomization to death from any cause, assessed for up to 2 years
  Defined as the proportion of patients alive after 2 years of follow-up time. Will be estimated and compared between the two arms using the Mantel-Haenszel test based (stratified by Eastern Cooperative Oncology Group [ECOG] performance status [PS] and lactate dehydrogenase [LDH]) based on two-sided overall type I error rate of 0.05 adjusting for two-interim analysis. Mantel-Haenszel test will compare the 2-year OS rates while controlling for the stratification factors. The difference in 2-year OS rates in arms A and B will be estimated and presented with 95% repeated confidence interval of Jennison-Turnbull. In addition, OS distribution will be estimated using the Kaplan-Meier method. The distribution of OS will be compared using the stratified log rank test. Hazard of OS will be estimated as a function of time in arm A and in arm B (as randomized in step 1 to arm A versus B) and presented graphically.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | The time from randomization to disease progression or death (whichever occurs first), assessed up to 5 years
  Evaluated based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Distribution will be estimated using the Kaplan-Meier method. PFS will be compared using the log-rank test.
Response rate | Up to 5 years
  According to RECIST 1.1. Response rates will be compared using the Mantel-Haenszel test (stratified by ECOG PS and LDH) test in arms A vs. B. Response rate for patients who are treated with ipilimumab/nivolumab before crossover (arm A) vs. for patients who were initially treated with dabrafenib/trametinib and crossed over to ipilimumab/nivolumab will be compared (arm D). Response rates will be compared using the Fisher's exact test.
Toxicity rate for individual adverse events (AEs) | Up to 5 years
  Will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.0. Compared using the chi-square of Fisher's exact test. Two-sided p-values will be reported for these comparisons.
Toxicity rate for categorized AEs | Up to 5 years
  Will be assessed using CTCAE v 4.0. Compared using the chi-square of Fisher's exact test. Two-sided p-values will be reported for these comparisons.
Toxicity rate for worst degree AEs | Up to 5 years
  Will be assessed using CTCAE v 4.0. Compared using the chi-square of Fisher's exact test. Two-sided p-values will be reported for these comparisons.

OTHER OUTCOMES:
Genetic characteristics | Baseline
  Genetic associations with immune-related adverse events (irAE) status will be assessed using Fisher's exact test, one-degree-of-freedom genotypic trend test or the two-degrees-of-freedom chi-squared test of independence at each individual SNP marker. Tests of association will be adjusted for age, sex, center or clinical protocol, and dose as well as American Joint Committee on Cancer stage, ulceration, performance status, LDH level, number of involved sites, BRAF mutation status (when available) and number of prior therapies using logistic regression modeling assuming an additive genetic model.
Immune-related adverse events (irAE) status | Up to 2 years
  Genetic associations with irAE status will be assessed using Fisher's exact test, one-degree-of-freedom genotypic trend test or the two-degrees-of-freedom chi-squared test of independence at each individual SNP marker. Tests of association will be adjusted for age, sex, center or clinical protocol, and dose as well as American Joint Committee on Cancer stage, ulceration, performance status, LDH level, number of involved sites, BRAF mutation status (when available) and number of prior therapies using logistic regression modeling assuming an additive genetic model.
Quality-adjusted time without symptoms of disease progression or toxicity of treatment (Q-TWIST) | Up to 2 years
  The restricted mean amount of time for each health state will be estimated using the Kaplan-Meier method, with time limit set at 2 years for computation of all restricted means. The mean amount of time for each health state and the average group utility scores will be summarized by initial treatment (i.e., arm A: ipilimumab + nivolumab [with subsequent dabrafenib + trametinib] vs. arm B: dabrafenib + trametinib [with subsequent ipilimumab + nivolumab]). The Q-TWiST subscore and the overall Q-TWiST score will then be reported by initial treatment. Differences between treatment groups in the mean Q-TWiST score (including the overall score and the subscore) will be calculated. For each score, a 95% confidence interval and two-sided P-value for testing the null hypothesis of no difference between treatment groups will be conducted using a Z-test (with normal approximation), with standard errors calculated by the bootstrap method.
Overall function | Up to 24 months from study entry
  Assessed using Patient-Reported Outcomes Measurement Information System (PROMIS) PROFILE-29. A log-normal survival model for analyzing longitudinal data which incorporates the non-ignorable censoring mechanism will be fitted for each short form T-score and pain intensity, separately, to assess initial treatment effect (i.e., arm A: ipilimumab + nivolumab [with subsequent dabrafenib + trametinib] vs. arm B: dabrafenib + trametinib [with subsequent ipilimumab + nivolumab]) on each function. To evaluate the effect of treatment sequence on patient function, each of the PROMIS short form T-score and pain intensity (with longitudinal data collected at baseline, 6-, 12-weeks, and 6-months after the initiation of treatment in each step) will be compared by treatment sequence for ipilimumab + nivolumab (arm A vs. D) and for dabrafenib + trametinib (arm B vs. C), using a log-normal survival model as described above.
Change in patient-reported symptoms | Baseline to up to 6 months after the initiation of treatment in each step
  Assessed using the Patient Reported Outcomes Common Terminology Criteria for Adverse Events. To evaluate the effect of treatment sequence on symptoms, summary statistics (frequency [N] and percentage [%]) will be reported with respect to presence, frequency and severity (if applicable) for each symptom by treatment sequence for ipilimumab + nivolumab (arm A vs. D), and for dabrafenib + trametinib (arm B vs. C) at baseline, 6-, 12-weeks, and 6-months after the initiation of the first treatment and the secondary treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Atkins, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (843):
- United States (843):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Adventist Health Cancer Care Center Chico, Chico, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Mills Health Center, San Mateo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - The Medical Center of Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - Straub Pearlridge Clinic, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Kendrick Colon and Rectal Center-Indianapolis, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - FMH James M Stockman Cancer Institute, Frederick, Maryland
  - Mercy Medical Center, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - New York Oncology Hematology PC - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Wake Forest Baptist Health - Hematology Oncology - Statesville, Statesville, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Cancer Survival Center - West, Knoxville, Tennessee
  - Thompson Oncology Group-Maryville, Maryville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Thompson Oncology Group-Oak Ridge, Oak Ridge, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] Atkins MB, Lee SJ, Chmielowski B, Tarhini AA, Cohen GI, Truong TG, Moon HH, Davar D, O'Rourke M, Stephenson JJ, Curti BD, Urba WJ, Brell JM, Funchain P, Kendra KL, Ikeguchi AP, Jaslowski A, Bane CL, Taylor MA, Bajaj M, Conry RM, Ellis RJ, Logan TF, Laudi N, Sosman JA, Crockett DG, Pecora AL, Okazaki IJ, Reganti S, Chandra S, Guild S, Chen HX, Streicher HZ, Wolchok JD, Ribas A, Kirkwood JM. Combination Dabrafenib and Trametinib Versus Combination Nivolumab and Ipilimumab for Patients With Advanced BRAF-Mutant Melanoma: The DREAMseq Trial-ECOG-ACRIN EA6134. J Clin Oncol. 2023 Jan 10;41(2):186-197. doi: 10.1200/JCO.22.01763. Epub 2022 Sep 27. PMID 36166727
- [Derived] Barker CA, Salama AK. New NCCN Guidelines for Uveal Melanoma and Treatment of Recurrent or Progressive Distant Metastatic Melanoma. J Natl Compr Canc Netw. 2018 May;16(5S):646-650. doi: 10.6004/jnccn.2018.0042. PMID 29784747